CLINICAL TRIAL: NCT03639727
Title: Cough in Eastern and Central Finland
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Heikki Koskela, Professor, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KUH5801136
Record Dates: First submitted 2018-08-09; First posted 2018-08-21 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Chronic Cough
Keywords: cough; cough provocation test; mannitol; citric acid
MeSH Terms: conditions — Chronic Cough; Cough

STUDY DESIGN:
Intervention Model Description: This study compares citric acid and mannitol bronchial challenges in their ability to separate chronic cough subjects from healthy subjects. There are no therapeutic interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citric acid aerosol bronchial challenge (Active Comparator): Inhaled citric acid aerosol. This study investigates the diagnostic accuracy of two cough provocation tests, one of which is citric acid aerosol challenge.
  Interventions: Diagnostic Test: Citric acid aerosol bronchial challenge
- Mannitol aerosol bronchial challenge (Active Comparator): Inhaled mannitol aerosol. This study investigates the diagnostic accuracy of two cough provocation tests, one of which is mannitol aerosol challenge.
  Interventions: Diagnostic Test: Mannitol aerosol bronchial challenge

INTERVENTIONS:
Diagnostic Test: Citric acid aerosol bronchial challenge — Inhalation challenge by citric acid aerosol to investigate the subject's cough sensitivity
  Arms: Citric acid aerosol bronchial challenge
Diagnostic Test: Mannitol aerosol bronchial challenge — Inhalation challenge by mannitol aerosol to investigate the subject's cough sensitivity
  Arms: Mannitol aerosol bronchial challenge

SUMMARY:
Comparison of citric acid and mannitol cough provocation tests among subjects with chronic cough and healthy volunteers.

DETAILED DESCRIPTION:
35 subjects with chronic cough plus 25 subjects without any cough will be asked to participate. The study consists of two visits in the outpatient clinic of Kuopio University Hospital, department of respiratory medicine, 2 - 7 days apart. They will fill in the Leicester Cough Questionnaire and undergo two different cough provocation tests, in random order: Mannitol test and citric acid test. If a chest x-ray has not been taken within 6 months, it will be taken.

ELIGIBILITY:
Inclusion Criteria, Chronic cough patients:

(both criteria must be fulfilled)

* presence of current chronic cough (> 8 weeks)
* Leicester Cough Questionnaire total score < 17

Inclusion criteria, healthy volunteers

* absence of any form of cough

Exclusion Criteria:

* age < 18 years
* any disability which would challenge the subject's ability to understand the purpose and methods of the study
* pregnancy
* breastfeeding
* current smoking or ex smoking more than 10 pack years
* any thoracic x-ray finding indicating urgent mediacal interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Receiver operator characteristic curves of the citric acid and the mannitol aerosol bronchial challenges | Within one week from the start of the study in each individual
  Receiver operator characteristic curve describes the ability of the bronchial challenge to separate the cough patients from healthy volunteers

SECONDARY OUTCOMES:
Leicester Cough Questionnaire total score | The first study day
  Measures cough-spesific quality of life. Range is 3 - 21 with low total score indicating poor cough-spesific quality of life. The three Leicester Cough Questionnaire subscales are added together to form the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Heikki O Koskela, MD, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pautola HVT, Koskela HO, Purokivi MK, Kaulamo JT, Latti AM. The prevalence and risk factors of respiratory symptoms in Finland: a comparative analysis. Eur Clin Respir J. 2025 Sep 25;12(1):2563395. doi: 10.1080/20018525.2025.2563395. eCollection 2025. PMID 41020184